CLINICAL TRIAL: NCT01952184
Title: Oocyte Survival After Vitrification in an Open or Closed Commercial Device: Study on Sibling Donor Oocytes.
Brief Title: Oocyte Survival After Vitrification in an Open or Closed Device With Closed Storage.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Neelke De Munck, MSc., Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/777
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Survival; Embryo Quality
Keywords: vitrification; oocyte; donor; open; closed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- closed vitrification with closed storage (Active Comparator): Half of the oocytes of every donor will be vitrified with the Cryo Bio Systems High Security vitrification (CBSvit HS) device; the standard device in our lab.
  Interventions: Device: CBSvit HS device
- open vitrification with closed storage (Experimental): Half of the oocytes of every donor will be vitrified with the Cryotop closed system (Cryotop SC).
  Interventions: Device: Cryotop SC device

INTERVENTIONS:
Device: CBSvit HS device — closed vitrification with closed storage
  Arms: closed vitrification with closed storage
Device: Cryotop SC device — open vitrification with closed storage
  Arms: open vitrification with closed storage

SUMMARY:
The survival rate (and embryo quality) of donor oocytes with two commercially available devices.

DETAILED DESCRIPTION:
Donor sibling oocytes will be vitrified with two commercially available devices. The first device is closed vitrification with closed storage and the second device is open vitrification with closed storage. Oocyte acceptors receive oocytes from both devices. With the increase in cooling rate generated by the open vitrification (second device), we expect to get an increase in survival rate of 10%. Besides this, embryo quality will be assessed with oocytes obtained from both devices.

ELIGIBILITY:
Inclusion Criteria:

* Donor: ≤36 years old on day of oocyte retrieval
* Donor: ≥ 6 mature oocytes

Exclusion Criteria:

* Donor: < 6 mature oocytes

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Survival rate | up to 6 days after every warming cycle
  The purpose is to assess the survival rate of donor oocytes with the two vitrification devices.

SECONDARY OUTCOMES:
Embryo development | up to 6 days after every warming cycle
  The purpose is to analyse the pre-implantation development of donor oocytes vitrified with two different devices.

CONTACTS AND LOCATIONS:
Overall Officials: Neelke De Munck, MSc., Principal Investigator — Centrum voor Reproductieve Geneeskunde, UZBrussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

REFERENCES:
- [Derived] De Munck N, Santos-Ribeiro S, Stoop D, Van de Velde H, Verheyen G. Open versus closed oocyte vitrification in an oocyte donation programme: a prospective randomized sibling oocyte study. Hum Reprod. 2016 Feb;31(2):377-84. doi: 10.1093/humrep/dev321. Epub 2016 Jan 2. PMID 26724798